CLINICAL TRIAL: NCT06128473
Title: Clinical Evaluation of the Safety and Efficacy of Yung Sheng 38% Color Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yung Sheng Optical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE-120901
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Contact Lenses, Hydrophilic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yung Sheng 38% color contact lens (Experimental)
  Interventions: Device: Soft Contact Lens

INTERVENTIONS:
Device: Soft Contact Lens — Vision Correction

SUMMARY:
This was a single group, open-label clinical study to assess the safety and efficacy of Yung Sheng 38% color contact lens for vision correction.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must sign the informed consent form.
2. The subject must be at least 20 years of age as of the date of evaluation for the study.
3. The subject must have a spherical prescription range between 0 to -12.00 diopters in each eye.
4. The subject must have manifest refraction Snellen visual acuities (VA) less than 0.8 in each naked eye.
5. The subject must have normal eyes, except ametropia.
6. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
7. The subject must appear able and willing to fill the daily card.

Exclusion Criteria:

1. The subjects who need to use ophthalmic medicine for therapy.
2. The subjects who have ocular or systemic allergies or disease that may interfere with contact lens wear.
3. The subjects who have any history of ocular surgery/injury within 8 weeks prior to enrollment.
4. The subjects who have clinically significant tear secretion abnormal.
5. The subjects who enrolled in another contact lens clinical trial within 30 days prior to enrolment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 71 (Actual)
Dates: Start 2013-06-18 (Actual); Primary Completion 2014-07-03 (Actual); Study Completion 2014-07-03 (Actual)

PRIMARY OUTCOMES:
The effectiveness of corrected visual acuity | 3 Months
  The visual acuity after contact lens correction should be more than or equal to 1.0 at the final visit for each subject. The percentage of successful contact lens correction of visual acuity should be more than 90 % among all subjects.

SECONDARY OUTCOMES:
Lens fitting (Lens position) | Day 1, 1 week, 2 weeks, 1 month, 2 months and 3 months
  Lens position should be "in the middle of eyes". The successful percentage among all subjects should be more than 80 %.
  Slit-lamp biomicroscopy will be assessed according to the approved study biomicroscopy CRF.
Lens fitting (Lens movement) | Day 1, 1 week, 2 weeks, 1 month, 2 months and 3 months
  Lens movement should be less than "1.5 mm". The successful percentage among all subjects should be more than 80 %.
  Slit-lamp biomicroscopy will be assessed according to the approved study biomicroscopy CRF.
Lens fitting (Lens edge) | Day 1, 1 week, 2 weeks, 1 month, 2 months and 3 months
  Lens edge should be normal after wearing. The successful percentage among all subjects should be more than 80 %.
  Slit-lamp biomicroscopy will be assessed according to the approved study biomicroscopy CRF.

OTHER OUTCOMES:
Safety evaluation | 12 weeks
  1. Incidence of adverse events;
  2. Incidence of serious adverse events;
  The safety endpoint in this evaluation is the rate of serious adverse reactions related to visual acuity loss as well as accompanying slit-lamp findings and other associated observations.
  [Time Frame: 12 weeks]

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Yu Tsai, PhD, Principal Investigator — China Medical University Hospital; Mei-Ling Peng, PhD, Principal Investigator — Chung Shan Medical University